CLINICAL TRIAL: NCT02000050
Title: Phase II Study of Up-front Chemotherapy and Neo-adjuvant Short-course Radiotherapy for Resectable Rectal Carcinoma
Brief Title: Phase II Study of Up-front Chemotherapy and Neo-adjuvant Short-course Radiotherapy for Resectable Rectal Carcinoma (COLORE)
Acronym: COLORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST154.01; 2013-000770-30 (EudraCT Number)
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Rectal Carcinoma
Keywords: resectable rectal cancer; up-front chemotherapy; neo-adjuvant short course radiotherapy; short course radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Folfox protocol; Radiotherapy, Intensity-Modulated; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): * Neoadjuvant therapy: FOLFOX4 2 cycles + Tomotherapy + FOLFOX4 2 cycles
  * Surgery
  * Adjuvant therapy: FOLFOX4 8 cycles
  * TME (Total Mesorectal Excision)
  Interventions: Drug: FOLFOX4; Radiation: Tomotherapy; Procedure: TME (Total Mesorectal Excision)

INTERVENTIONS:
Drug: FOLFOX4 — FOLFOX4
Radiation: Tomotherapy — Tomotherapy
Procedure: TME (Total Mesorectal Excision) — TME (Total Mesorectal Excision)
  Other Names: surgery

SUMMARY:
Phase II study of up-front chemotherapy and neo-adjuvant shortcourse radiotherapy for resectable rectal carcinoma.

Study Design: Phase II, open-label, single-arm, multi-centre study.

STUDY PRODUCT,DOSE,ROUTE,REGIMEN AND DURATION OF ADMINISTRATION:

1. Neoadjuvant Treatment (pre-operative chemo-radiotherapy regimen):

   FOLFOX4* 2 cycles (WK1+WK3) - Tomotherapy** (WK5) - FOLFOX4* 2 cycles (WK7+WK9)

   * Oxaliplatin 85 mg/m2 iv: day 1 Levofolinate 100 mg/m2 iv: day 1-2 5-fluorouracil 400 mg/m2 iv in bolus and 600 mg/m2 iv infusion over 22h: day 1-2 Every cycle will last 2 weeks (approximately 48 hours of treatment infusion and 12 days of rest).

   ** 25 Gy in 5 consecutive fractions, one fraction per day in 5 days on CTV (Clinical Target Volume) at the isodose of the 95% of the total dose. The treatment plan will be elaborated at the work-station dedicated to the Helicoidal Tomotherapy. The treatment could be planned also with linear accelerator with IGRT-IMRT technique or VMAT technique.
2. Restaging (week 11)
3. Surgery (week 12-16) with Total Mesorectal Excision (TME)
4. End Of Treatment (week 16-32)
5. Adjuvant therapy (The maximum interval between surgery and start of adjuvant therapy should be 8 weeks):
6. FOLFOX4* 8 cycles (every 2 weeks)

Study Duration: about 5 years. Enrollment period: 36 months. Treatment period: about 8 months. Follow-up: 1 year.

NUMBER OF SUBJECTs:

· Step A: a maximum of 6 patients. 6 evaluable patients are needed to assess toxicity. If 1 toxicity resulting in discontinuation of treatment will be observed in 6 patients, the treatment can be considered safe (with a confidence > 90%).

If 2 or more toxicity resulting in discontinuation of treatment on 6 patients, the study will be stopped because not safe and another type of radiotherapy schedule must be designed.

· Step B: a total of 50 patients is required to be recruited in 2 years (including patients enrolled in Step A).

The goal is to achieve a proportion of at least 15% of patients with a complete pathological response with the new radiochemotherapeutic treatment.

DETAILED DESCRIPTION:
Title: Phase II study of up-front chemotherapy and neo-adjuvant shortcourse radiotherapy for resectable rectal carcinoma.

Short Title/Acronym: COLORE

Protocol Code: IRST154.01

Phase: 2

Study Design: Phase II, open-label, single-arm, multi-centre study.

STUDY PRODUCT,DOSE,ROUTE,REGIMEN AND DURATION OF ADMINISTRATION:

1. Neoadjuvant Treatment (pre-operative chemo-radiotherapy regimen):

   FOLFOX4* 2 cycles (WK1+WK3) - Tomotherapy** (WK5) - FOLFOX4* 2 cycles (WK7+WK9)

   * Oxaliplatin 85 mg/m2 iv: day 1 Levofolinate 100 mg/m2 iv: day 1-2 5-fluorouracil 400 mg/m2 iv in bolus and 600 mg/m2 iv infusion over 22h: day 1-2 Every cycle will last 2 weeks (approximately 48 hours of treatment infusion and 12 days of rest).

   ** 25 Gy in 5 consecutive fractions, one fraction per day in 5 days on CTV (Clinical Target Volume) at the isodose of the 95% of the total dose. The treatment plan will be elaborated at the work-station dedicated to the Helicoidal Tomotherapy. The treatment could be planned also with linear accelerator with IGRT-IMRT technique or VMAT technique.
2. Restaging (week 11)
3. Surgery (week 12-16) with Total Mesorectal Excision (TME)
4. End Of Treatment (week 16-32)
5. Adjuvant therapy (The maximum interval between surgery and start of adjuvant therapy should be 8 weeks):
6. FOLFOX4* 8 cycles (every 2 weeks)

Study Duration: about 5 years. Enrollment period: 36 months. Treatment period: about 8 months. Follow-up: 1 year.

OBJECTIVES

Primary objectives:

Step A: to evaluate the feasibility and safety of the chemoradiotherapy regimen.

Step B: to evaluate the proportion of patients with pathological complete remission after combined radio-chemotherapy.

Secondary objectives (of Step B):

* To evaluate the safety of the neo-adjuvant treatment
* To determine pathological down-staging
* To evaluate the rate of R0 resection
* To evaluate the sphincter saving resection rate
* To evaluate median disease free survival and overall survival
* To evaluate the correlation between biomarker, pathological response and outcome (auxiliary\subsidiary Biological Study)

NUMBER OF SUBJECT:

· Step A: a maximum of 6 patients. 6 evaluable patients are needed to assess toxicity. If 1 toxicity resulting in discontinuation of treatment will be observed in 6 patients, the treatment can be considered safe (with a confidence > 90%).

If 2 or more toxicity resulting in discontinuation of treatment on 6 patients, the study will be stopped because not safe and another type of radiotherapy schedule must be designed.

· Step B: a total of 50 patients is required to be recruited in 2 years (including patients enrolled in Step A).

The goal is to achieve a proportion of at least 15% of patients with a complete pathological response with the new radiochemotherapeutic treatment.

STATISTICAL METHODOLOGY:

The primary analysis will be performed on the ITT (Intention-To-Treat) population, while the secondary analysis will be conducted on the PP (Per Protocol) population.

The number and percentage of treated patients undergoing grade 1 to 4 adverse events (CTC-AE, version 4.0) will be tabulated in the ITT and PP population. No statistical inference will be performed.

Step A: Patients, tumor characteristics and toxicity events observed will be described.

Step B: The proportion of patients with pathological Complete Response will be calculated. Safety profile will be analyzed. OS (Overall Survival) and DFS (Disease Free Survival) will be estimated with Kaplan-Meier method (Kaplan El, Meier P., J Am Stat Assoc 1958).

No interim analysis will be performed. The 95% confidence intervals should also be provided.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed diagnosis of adenocarcinoma of the mid-low rectum (within 12 cm from the anal verge)
2. Stage: lowT2N0, T2N+M0, T3-4 N-/+M0 (N+ = ≥ 3 nodes >0,5 cm diameter or ≥ 1 nodes > 1 cm diameter)
3. Age ≥18 and ≤ 80 years
4. ECOG performance status 0-1
5. Patients must have normal organ and marrow function as defined below:

   1. - Leukocytes ≥ 3,000/mL
   2. - Absolute neutrophil count ≥ 1,500/mL
   3. - Platelets ≥ 100,000/mL
   4. - Total bilirubin ≤ 1.5 X ULN
   5. - AST (SGOT)/ALT (SGPT) ≤ 2.5 X ULN
   6. - Creatinine ≤ 1.5 X ULN
6. Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
7. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Metastatic disease
2. Patients who have had any chemotherapy or radiotherapy prior to entering the study
3. Acute or sub-acute gastrointestinal occlusion
4. Participation in another clinical trial, with any investigational agent within 30 days prior the study screening
5. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma, superficial bladder tumor and in situ carcinoma of the uterine cervix)
6. History of allergic reactions attributed to compounds of similar chemical or biological composition to drugs used in the study
7. Uncontrolled concomitant illness, including but not limited to: ongoing or active infections; congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance to study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-10-11 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Toxicity events | 15 months
  6 evaluable patients are needed to assess toxicity. If one toxicity resulting in discontinuation of treatment will be observed in 6 patients, we can conclude that the true probability of toxicity is less than 45% with a confidence >90% and the treatment can be considered safe. If 2 or more toxicity resulting in discontinuation of treatment on 6 patients we can conclude that the true probability of toxicity is greater than 10% with a confidence >90%, and the study will be stopped because not safe and another type of radiotherapy schedule must be designed.
The Simon optimal two-stage design (Richard Simon, Controlled Clinical Trials 1989) | 15 months
  It's a two-stage design that use for P1(the proportion of pCR with the new radio-chemotherapeutic treatment) - P0 (the expected proportion of pCR) =0.15. It's used to understand if a treatment is active or not.
Complete pathological response (pCR) | 3 years
  According to pathological response criteria, a total regression is considered a complete response. This parameter is used to understand if a treatment is active or not ( if at least 7 patients out of 50 enrolled will achieve a pCR, the treatment could be considered active).

SECONDARY OUTCOMES:
Objective tumor response rate (ORR) | 5 years
  It is the proportion of the intention-to-treat (ITT) population showing a complete or partial response, if confirmed ≥ 4 weeks later.
  It will be assessed using RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
Pathological Downstaging Rate | 5 years
  The proportion of subjects with an improved histopathological response by one or more grade relative to baseline following rectal surgery with Total Mesorectal Excision (TME).
Disease-free survival time (DFS) | 5 years
  The time from enrolment date to date of first observed progression, relapse or death.
Overall survival time (OS) | 5 years
  Time from enrolment to the date of death.
Intention-to-treat (ITT) population | 5 years
  The population of all enrolled patients with baseline assessment of disease, receiving 2 cycles of treatment of FOLFOX4 and at least 1 day of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Passardi, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (2):
- Italy (2):
  - UO Oncologia Medica IRCCS IRST, Meldola, FC
  - Oncologia Medica PO RAVENNA; FAENZA; LUGO, Ravenna, RA

REFERENCES:
- [Result] Passardi A, Rapposelli IG, Scarpi E, Neri E, Parisi E, Ghigi G, Ercolani G, Avanzolini A, Cavaliere D, Rudnas B, Valgiusti M, Barone D, Ferroni F, Frassineti GL, Romeo A. Neoadjuvant treatment (FOLFOX4 plus hypofractionated tomotherapy) for patients with locally advanced rectal cancer: a multicenter phase II trial. Ther Adv Med Oncol. 2020 Dec 8;12:1758835920977139. doi: 10.1177/1758835920977139. eCollection 2020. PMID 33343722